CLINICAL TRIAL: NCT06869850
Title: MFGM-EnhaNceD RUTF for Children With SAM
Brief Title: Milk Fat Globule Membrane-Enhanced RUTF for Children With Severe Acute Malnutrition
Acronym: MEND-SAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Project Peanut Butter (Other); Ministry of Health and Sanitation, Sierra Leone (Other Government); Arla Food Ingredients Group P/S (Unknown); The Danish Dairy Research Foundation, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202503015
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Severe Acute Malnutrition; Cognitive Impairment; Kwashiorkor; Severe Wasting
Keywords: severe acute malnutrition; severe wasting; kwashiorkor; milk fat globule membrane; neurodevelopment; phospholipids; ganglioside; dairy fat; malawi developmental assessment tool; Sierra Leone; ready-to-use therapeutic food
MeSH Terms: conditions — Severe Acute Malnutrition; Cognitive Dysfunction; Kwashiorkor; Cachexia | interventions — Amoxicillin; Sulfadoxine; Pyrimethamine

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MFGM-RUTF (Milk fat globule membrane ready-to-use therapeutic food) (Experimental): One sachet contains 92g of MFGM-RUTF. During SAM treatment, each participant will be given sufficient MFGM-RUTF to consume 2 sachets per day, which will provide approximately 1000 calories, 27g of protein, 63g of fat, and over 1 RDA of micronutrients.
  Interventions: Dietary Supplement: MFGM-RUTF (milk fat globule membrane ready-to-use therapeutic food); Drug: Amoxicillin; Drug: Sulfadoxine (12.5 mg)/Pyrimethamine (250 mg)
- S-RUTF (standard ready-to-use therapeutic food) (Active Comparator): One sachet contains 92g of S-RUTF. During SAM treatment, each participant will be given sufficient S-RUTF to consume 2 sachets per day, which will provide approximately 1000 calories, 27g of protein, 60g of fat, and over 1 RDA of micronutrients.
  Interventions: Dietary Supplement: S-RUTF (standard ready-to-use therapeutic food); Drug: Amoxicillin; Drug: Sulfadoxine (12.5 mg)/Pyrimethamine (250 mg)

INTERVENTIONS:
Dietary Supplement: MFGM-RUTF (milk fat globule membrane ready-to-use therapeutic food) — MFGM whey protein/fat concentrate powder used in place of skim milk powder in peanut paste-based ready-to-use therapeutic food meeting Codex Alimentarius specifications. There will be 10g of MFGM-containing whey protein/fat concentrate powder per 100g of MFGM-RUTF. Other ingredients and amounts per 100g: 9.5g rice flour, 5g whey permeate, 18.5g palm oil, 31g peanut paste, 22.1g sugar, 2.9g micronutrient mix, 1g fish oil.
  Arms: MFGM-RUTF (Milk fat globule membrane ready-to-use therapeutic food)
Dietary Supplement: S-RUTF (standard ready-to-use therapeutic food) — Standard peanut paste-based ready-to-use therapeutic food made with skim milk powder meeting Codex Alimentarius specifications. This RUTF is modeled on the most widely used recipe worldwide, containing per 100g: 19.5g skim milk powder, 9.3g palm oil, 7g canola oil, 31.3g peanut paste, 28g sugar, 1g soy flakes, 1g hydrogenated vegetable oil, and 2.9g micronutrient mix.
  Arms: S-RUTF (standard ready-to-use therapeutic food)
Drug: Amoxicillin — Oral amoxicillin tablets twice per day for 7 days dosed based on weight
Drug: Sulfadoxine (12.5 mg)/Pyrimethamine (250 mg) — Malaria chemoprophylaxis, dosed by weight, to be given every month during SAM treatment

SUMMARY:
The goal of this clinical trial is to test the use of milk fat globule membrane (MFGM) in ready-to-use therapeutic food (RUTF) in children with severe acute malnutrition in Sierra Leone. The main questions it aims to answer are:

* Will the inclusion of MFGM in RUTF for 6-59-month-old Sierra Leonean children with severe acute malnutrition improve their neurodevelopment?
* Will the inclusion of MFGM in RUTF for 6-59-month-old Sierra Leonean children with severe acute malnutrition reduce its worst consequences: death, hospitalization, and remaining severely malnourished despite treatment?

Researchers will compare the MFGM-containing RUTF to standard RUTF, which contains skim milk powder.

Participants will:

* undergo measurement of length, weight, mid-upper arm circumference, and nutritional edema assessment every two weeks during severe malnutrition treatment
* be treated with either MFGM-RUTF or standard RUTF at a dose of 2 sachets per day for up to 12 weeks
* undergo neurodevelopmental testing using the Malawi Developmental Assessment Tool at the end of SAM treatment and 6 months later
* a subset of participants will undergo blood spot collection and stool sample collection

DETAILED DESCRIPTION:
Globally, approximately 15 million children are suffering from severe acute malnutrition (SAM) at any one time, a number that has not declined in recent decades despite significant technological advancements in agriculture and food science. SAM is a condition of total-body depletion of the nutrients required for health and development; without treatment, 50% of affected children will die. Whereas historically children with SAM were admitted to and treated within hospitals, the advent of ready-to-use therapeutic food (RUTF) and community-based management of acute malnutrition revolutionized SAM care by allowing it to occur safely and successfully by the child's caregiver in their own home.

RUTF was designed to provide the nutrients required for physical recovery in a safe, palatable format. It is equal parts peanut paste, sugar, vegetable oil, and skim milk powder, with added micronutrients and emulsifier. At inception, attention was not specifically paid to how RUTF's composition might impact neurodevelopmental recovery in children with SAM. Research over the past decade has revealed that even following successful treatment with RUTF, children diagnosed with SAM still score 1-3 standard deviations below age-based expectations on neurodevelopmental tests. This suggests that the nutrient profile of standard RUTF is not sufficient to recover the developmental damage incurred by SAM.

Recently, progress has been made toward improving the developmental trajectory of children with SAM by altering RUTF. A randomized, blinded trial in Malawi including 2,500 children with SAM showed that improving the polyunsaturated fatty acid (PUFA) profile of RUTF by reducing linoleic acid and adding docosahexaenoic acid (DHA) yields superior neurodevelopment 6 months after treatment, by 0.19 standard deviations on a standardized, culturally adapted neurodevelopmental test. This demonstrates that neurodevelopmental recovery in SAM is sensitive to the lipid profile of RUTF. Despite the benefits of improved PUFA RUTF, however, children with SAM remained 1 standard deviation below expectations in neurodevelopment.

The milk fat globule membrane (MFGM) in mammalian milk contains a host of nutrients and bioactive compounds supportive of physical health and brain development. Bovine MFGM added to infant formula has been tested in several clinical trials and has demonstrated a reduction in infectious episodes, such as diarrhea and ear infections, as well as improvement in cognitive development, compared with infant formula not containing MFGM. In these trials and others, MFGM has been shown to be safe and well-tolerated. Currently, RUTF contains skim milk powder as its high-quality protein source, and peanut and vegetable oils as the primary sources of fat. These vegetable fat sources are deficient in the lipids provided by MFGM: sphingolipids, cholesterol, and other phospholipids such as phosphatidylcholine and phosphatidylethanolamine, all of which play roles in brain development. It is possible that the lipids contained in MFGM may further support neurodevelopmental recovery in SAM children.

By acting as a natural emulsifier, MFGM also offers a food formulation advantage that is relevant to children with SAM. Animal model studies have demonstrated that emulsifiers can compromise the gut barrier. Children with SAM have damaged small intestinal barrier function, which can lead to translocation of gut bacteria and resulting systemic infection. As RUTF will compose nearly 100% of a child's intake for the duration of treatment - up to 3 months - it is possible that inclusion of emulsifier may impede gut healing and recovery. Considering this concern, the Manary lab ran a clinical trial in 2018-2019 testing a novel formulation of RUTF designed with oat in place of some skim milk powder and peanut, and without hydrogenated vegetable oil (standard emulsifier), because oat acts as a natural emulsifier. In this trial, children with SAM receiving the oat-RUTF had 10% absolute higher recovery and a 33% relative reduction in the worst SAM outcomes (death, hospitalization, or remaining severely malnourished). Like oat, MFGM in RUTF allows for omission of emulsifier and may yield similar benefits.

Given (1) the repeated finding that adding MFGM to infant formulas improves neurodevelopment, (2) the impaired neurodevelopment of children with SAM, (3) the current RUTF formulation lacking neuro-supportive fats provided by MFGM, (4) MFGM's natural activity as an emulsifier, and (5), the reality that RUTF provides the sole source of nutrition for children with SAM, it is plausible that adding this high-quality source of lipids and protein to RUTF may also benefit children with SAM in both immediate and long-term physical and cognitive recovery.

This will be an individually randomized, investigator/outcomes assessors-blinded, controlled clinical trial designed to determine if treatment of severely malnourished Sierra Leonean children 6-59-months of age with an RUTF made with MFGM-containing whey protein/fat concentrate will (1) improve neurodevelopment and (2) reduce a composite of poor SAM outcomes (death, hospitalization, remaining severely malnourished), compared with standard RUTF (S-RUTF). This trial will be conducted at 20 rural sites in Sierra Leone. 1600 children will be randomized 1:1 to receive 2 sachets per day of either MFGM-RUTF or S-RUTF. Children will receive their allocated RUTF and return to clinic fortnightly for repeat anthropometric measurements, illness questions, and to receive more RUTF until they achieve a clinical outcome or for a maximum of 12 weeks, at which point they will undergo Malawi Developmental Assessment Tool (MDAT) testing. Participants will be asked to return to clinic 6 (5-7) months later for MDAT testing, the global z-score from which will be the trial's co-primary outcome. A subset of participants will undergo blood spot and/or stool sample collection at the end of SAM treatment.

ELIGIBILITY:
Inclusion Criteria:

* 6-59 months of age
* Reside within the catchment area of a participating clinic
* mid-upper arm circumference < 11.5 cm and/or weight-for-length z-score < -3 and/or presence of bilateral pedal pitting edema
* willingness to comply with all study procedures and availability for the duration of the study, including no plan to move from the catchment area of a participating clinic

Exclusion Criteria:

* Features of complicated SAM: inability to tolerate a 30 g test dose of RUTF, breathing difficulties, mental status changes, sepsis, diarrhea with severe dehydration, and/or physician/nursing clinical assessment that the child needs immediate hospitalization
* Participation in a separate therapeutic feeding program within the past month
* Known allergy to study food ingredient (peanut, milk, fish)
* Clinically evident developmental delay (most often determined based on research nursing assessment of physical appearance, movement, and informal discussion with caregiver)
* Presence of a chronic severe medical condition (other than tuberculosis and HIV), such as congenital heart disease

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1600 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Malawi Developmental Assessment Tool global z-score | 6 (5-7) months after SAM treatment completion
  Age-standardized score, -6 to +6, higher scores are better
Composite of poor severe acute malnutrition treatment outcomes | 2-12 weeks of therapeutic feeding
  This composite outcome will include death, hospitalization, and remaining severely malnourished despite 12 weeks of treatment

SECONDARY OUTCOMES:
Malawi Developmental Assessment Tool gross motor domain z-score | 6 (5-7) months after SAM treatment completion
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool fine motor domain z-score | 6 (5-7) months after SAM treatment completion
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool language domain z-score | 6 (5-7) months after SAM treatment completion
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool social-emotional domain z-score | 6 (5-7) months after SAM treatment completion
  Age-standardized score, -6 to +6, higher scores are better
Remaining severely malnourished at end of SAM treatment | 12 weeks of therapeutic feeding
  For MUAC enrollment: MUAC < 11.5 cm For WLZ enrollment: WLZ < -3 For enrollment by both MUAC and WLZ: either remaining in SAM range For nutritional edema enrollment: continued edema
Death during SAM treatment | 2-12 weeks of therapeutic feeding
  As per caregiver/family report
Hospitalization during SAM treatment | 2-12 weeks of therapeutic feeding
  Participant determined to require hospitalization. Determination may be made by caregiver/family, government health workers, or may be recommended by trial staff for clinical decompensation.
Graduation from SAM treatment | 2-12 weeks of therapeutic feeding
  For MUAC enrollment: MUAC ≥ 12.5cm For WLZ enrollment: WLZ > -2 based on enrollment length For MUAC and WLZ enrollment: may meet either For edema enrollment: resolution of edema, with at least 4 weeks treatment
Malawi Developmental Assessment Tool global z-score | Within 1 month of SAM treatment completion
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool gross motor domain z-score | Within 1 month of SAM treatment completion
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool fine motor domain z-score | Within 1 month of SAM treatment completion
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool language domain z-score | Within 1 month of SAM treatment completion
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool social-emotional domain z-score | Within 1 month of SAM treatment completion
  Age-standardized score, -6 to +6, higher scores are better
Rate of weight change | Across initial 4 weeks of therapeutic feeding, or 2 weeks if graduate after 2 weeks
  g / kg / day
Rate of length change | Across 2-12 weeks of therapeutic feeding
  mm / week
Rate of mid-upper arm circumference change | Across 2-12 weeks of therapeutic feeding
  mm / week
Rate of change in length-for-age z-score across entire follow-up | 7-10 months (2-12 weeks of therapeutic feeding, 5-7 months of follow-up thereafter)
  Difference in LAZ at final visit and initial visit divided by time months transpired
Diarrhea incidence during SAM treatment | 2-12 weeks of therapeutic feeding
  Caregiver report of participant diarrhea (>2 loose stools per day) during SAM treatment
Fever incidence during SAM treatment | 2-12 weeks of therapeutic feeding
  Caregiver report of participant fever during SAM treatment
Plasma DHA status at end of SAM treatment | Collected after 2-12 weeks of therapeutic feeding
  Blood spot DHA % total fatty acids in subset of participants at end of therapeutic feeding
Fecal host mRNA transcripts as markers of environmental enteric dysfunction at end of SAM treatment | Collected after 2-12 weeks of therapeutic feeding
  CD53, CDX1, HLA-DRA, TNF, S100A8, MUC12, and REG1A
Malawi Developmental Assessment Tool global z-score trajectory | 6 (5-7) months after SAM treatment completion
  Change in MDAT global z-score between initial test and final test

OTHER OUTCOMES:
Malawi Developmental Assessment Tool global z-score in sub-groups | 6 (5-7) months after SAM outcome
  Age-standardized score, -6 to +6, higher scores are better. Will be tested in subgroups based on SAM treatment outcome (graduation vs. other), age at enrollment, and sex
Malawi Developmental Assessment Tool global z-score in sub-groups | Within 1 month of SAM treatment completion
  Age-standardized score, -6 to +6, higher scores are better. Will be tested in subgroups based on SAM treatment outcome (graduation vs. other), age at enrollment, and sex
Composite of poor severe acute malnutrition treatment outcomes | 2-12 weeks of therapeutic feeding
  This composite outcome will include death, hospitalization, and remaining severely malnourished despite 12 weeks of treatment. This will be tested in subgroups by age at enrollment, sex, and enrollment criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Manary, MD, Principal Investigator — Washington University School of Medicine; Kevin B Stephenson, MD, Principal Investigator — Washington University School of Medicine; Indi Trehan, MD, MPH, Study Director — University of Washington
Locations (10):
- Sierra Leone (10):
  - Bandajuma, Bandajuma, Pujehun
  - Bandasuma, Bandasuma, Pujehun
  - Bendu Malen, Bendu Malen, Pujehun
  - Gbondapi, Gbondapi, Pujehun
  - Jendema, Jendema, Pujehun
  - Potoru, Potoru, Pujehun
  - Sahn Malen, Sahn Malen, Pujehun
  - Taninahun, Taninahun, Pujehun
  - Zimmi, Zimmi, Pujehun
  - Static, Pujehun

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 12 months of primary publication